CLINICAL TRIAL: NCT03294187
Title: Encouragement-induced Movement Therapy in Daily Life - a Randomized Controlled, Assessor-blinded Multi-center Trial in Stroke Patients With a Unilateral Hemiparesis, Using a Wrist-worn Tracking and Feedback Device
Brief Title: Encouragement-induced Movement Therapy in Daily Life
Acronym: ISEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Tyromotion AG (Unknown); Swiss Federal Institute of Technology in Zurich (ETH Zurich) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-00948
Record Dates: First submitted 2017-09-12; First posted 2017-09-26 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Stroke
Keywords: Upper Extremity; Feedback; Rehabilitation; Randomized Controlled Trial
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monitoring and Feedback (Experimental): Subjects will use two wrist-worn wearables over a period of 6 weeks. Patients will receive multimodal (vibrotactile and visual) feedback.
  Interventions: Device: Wrist-worn wearables
- Monitoring (Placebo Comparator): Study subjects will use identical devices over a period of 6 weeks. Patients will *not* receive multimodal feedback.
  Interventions: Device: Wrist-worn wearables

INTERVENTIONS:
Device: Wrist-worn wearables — See arm/group description.

SUMMARY:
Stroke places a major burden on health care and society. It often leads to a hemiparesis. Intensive stroke rehabilitation speeds up recovery. In daily practice, the financial and/or human resources to provide this intensive rehabilitation are often lacking. Applying modern-day tracking and feedback technology to encourage a self-administered, context specific training is expected to offer significant potential to increase intensity of practice. Up until now, there has been no randomized trial examining the effect of such an intervention on daily arm usage.

The primary objective of this study is to determine the effect of wearing an activity tracking and multimodal feedback device for six weeks on self-reported daily life use of the paretic arm after stroke, when compared to control group stroke subjects wearing a hardware-wise identical sham device providing no feedback. The secondary aim is to examine compliance to use the device and the quantitative, qualitative and functional improvement of the paretic arm. It is hypothesized that participants in the experimental group show a higher change in self-reported daily life use of the paretic arm when compared to the control group both post intervention and at 6-week follow-up.

ISEAR is a multicenter, assessor-blinded randomized controlled trial of 62 subjects beyond the first 3 months poststroke.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age with unilateral stroke and residual hemiparesis leading to a decrease of arm function after completion of all inpatient rehabilitation (at least 90 days post stroke)
* Ability to lift arm against gravity (>30 degrees flexion or abduction)
* Ability to don/doff the devices on both wrists independently or with assistance of a caregiver
* Ability to give informed consent as documented by signature

Exclusion Criteria:

* Major untreated depression
* Severe cognitive impairment
* Suffering from comprehensive aphasia
* Severely impaired sensation (unable to feel a soft touch on the dorsal side of their paretic wrist with closed eyes)
* Other major comorbidities (e.g., cardiopulmonary disease, renal failure, hepatic dysfunction, orthopedic disorders, etc.)
* Expected hospitalization during study period
* Known intolerance to device material
* Known or suspected non-compliance, drug or alcohol abuse
* The investigator, his/her family members, employees, and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Motor Activity Log - 14, Amount of Use sub scale | Post-intervention (6 weeks)
  Self-reported amount of upper limb use in daily life

SECONDARY OUTCOMES:
Fugl-Meyer Assessment, Upper Extremity sub scale | Post-intervention (6 weeks)
  Upper limb motor function
Fugl-Meyer Assessment, Upper Extremity sub scale | Follow-up (12 weeks)
  Upper limb motor function
Action Research Arm Test | Post-intervention (6 weeks)
  Upper limb capacity
Action Research Arm Test | Follow-up (12 weeks)
  Upper limb capacity
Modified Rankin Scale | Post-intervention (6 weeks)
  Global Disability
Modified Rankin Scale | Follow-up (12 weeks)
  Global Disability
EuroQol five dimensions five levels questionnaire | Post-intervention (6 weeks)
  Quality of Life
EuroQol five dimensions five levels questionnaire | Follow-up (12 weeks)
  Quality of Life
Motor Activity Log - 14, Quality of Movement sub scale | Post-intervention (6 weeks)
  Self-reported quality of upper limb use in daily life
Motor Activity Log - 14, Quality of Movement sub scale | Follow-up (12 weeks)
  Self-reported quality of upper limb use in daily life
Motor Activity Log - 14, Amount of Use sub scale | Follow-up (12 weeks)
  Self-reported amount of upper limb use in daily life

OTHER OUTCOMES:
Global Rating of Perceived Change | Post-intervention (6 weeks)
Global Rating of Perceived Change | Follow-up (12 weeks)
Concomitant movement therapy | Post-intervention (6 weeks)
  Time spend at Movement therapy (e.g., Physiotherapy, Occupational therapy)
Concomitant movement therapy | Follow-up (12 weeks)
Adverse Events | Baseline (0 week)
  Safety
Adverse Events | Post-intervention (6 weeks)
  Safety
Adverse Events | Follow-up (12 weeks)
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Andreas R Luft, Prof. MD, Principal Investigator — University of Zurich
Locations (3):
- Switzerland (3):
  - Cereneo, Center For Neurology and Rehabilitation, Vitznau
  - Zürcher RehaZentrum Wald, Wald
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mayrhuber L, Andres SD, Legrand ML, Luft AR, Ryser F, Gassert R, Veerbeek JM, Duinen JV, Schwarz A, Franinovic K, Rickert C, Schkommodau E, O Held JP, Easthope CA, Lambercy O. Encouraging arm use in stroke survivors: the impact of smart reminders during a home-based intervention. J Neuroeng Rehabil. 2024 Dec 21;21(1):220. doi: 10.1186/s12984-024-01527-2. PMID 39707385
- [Derived] Held JPO, Luft AR, Veerbeek JM. Encouragement-Induced Real-World Upper Limb Use after Stroke by a Tracking and Feedback Device: A Study Protocol for a Multi-Center, Assessor-Blinded, Randomized Controlled Trial. Front Neurol. 2018 Jan 25;9:13. doi: 10.3389/fneur.2018.00013. eCollection 2018. PMID 29422881